CLINICAL TRIAL: NCT05755880
Title: Effect of Addition of Single Low Dose Dexamethasone to Local Anesthetic in Caudal Analgesia on Healing Process After Pediatric and Adolescent Orthopaedic Surgery
Brief Title: Low Dose Dexamethasone to Local Anesthetic in Caudal Analgesia on Healing Process After Orthopaedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaaeldin Mohamed Abdelhafez, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDDLA
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (No Intervention)
- Dexamethason (Active Comparator)
  Interventions: Procedure: Intrathecal dexamethason

INTERVENTIONS:
Procedure: Intrathecal dexamethason — After general anesthesia intrathecal dexamthasone will be added
  Arms: Dexamethason

SUMMARY:
Addition of dexamethasone to local anesthetics infiltration has been proven to augment postoperative analgesia, prolongs anesthesia time and sometimes reduces the needed dose of local anesthetics and consequently, decreases their side effects and enhances early ambulation and hospital discharge (mainly due to decreased need for opioid use

DETAILED DESCRIPTION:
Long-term corticosteroids prescribing was associated with many adverse effects, as increased skin pigmentation, lowering immunity (catching opportunistic infections like herpes zoster, candida and cutaneous abscesses or even flaring localized infections), resistant hyperglycemia, renal impairment, hypertension, impaired healing, thinning skin that bruises easily, adrenal gland suppression, facial erythema, stria, acne, mild hirsutism, blurring vision, muscle weakness, glaucoma, cataract, thinning of hair, osteoporosis, and psychiatric disturbances (including mood fluctuations, depression or manic disorders).

Localized infection at site of injection is a known logical absolute contraindication for any injection including corticosteroids due to fearing of flaring of infection. Also, there is no single published article discussing an infection due to corticosteroids injection as an adjuvant to local anesthetics as it is always explained by inadequate aseptic technique performance.

In this study we will search if there is a role for corticosteroids in delaying healing process after orthopedic surgery. And compare the incidence of postoperative infection after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 1month up to 18 years old 2. Orthopaedic surgeries with average time up to one hour 3. Traumatic and orthopaedic indications for surgery

Exclusion Criteria:

1- Open fractures 2. Infected surgery 3. Hypersensitivity to dexamethasone 4. Bad nutritional conditions as Marasmus, Cerebral palsy and Kwashiorkor

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 30 minutes after recovery
  Visual analogue scale (VAS) for assessment of children's pain perception

REFERENCES:
- [Background] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428